CLINICAL TRIAL: NCT07176208
Title: Dose Ranging Clinical Study to Evaluate the Effects of Oral Delta-9-tetrahydrocannabinol (Δ9-THC) With and Without Alcohol on Perception and Driving Performance in Healthy Adults
Brief Title: Clinical Study to Evaluate the Effects of Oral Delta-9-tetrahydrocannabinol (Δ9-THC) With and Without Alcohol on Perception and Driving Performance in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Food and Drug Administration (FDA) (U.S. Federal Agency)
Collaborators: Spaulding Clinical Research LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: SCR-017
Record Dates: First submitted 2025-09-08; First posted 2025-09-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cannabis, Drug Effects; Driving Performance
Keywords: delta-9-tetrahydrocannabinol; Cannabis drug effects; Driving Performance; Subjective Perception; THC and alcohol
MeSH Terms: conditions — Marijuana Abuse | interventions — Dronabinol; Ethanol

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, 6-period crossover study in 48 healthy adult volunteers. This study has six 1-day treatment periods with at least 7-day washout between each period.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study will be double-blind, and the blind will be maintained through a randomization schedule held by the dispensing pharmacist. The pharmacist (and designated staff member responsible for confirmation of study drug dose and measurement of blood alcohol concentration) will be unblinded to subject treatment assignment; however, the pharmacist and any unblinded staff will not perform any study procedures other than study drug preparation, and dispensing, and measuring blood alcohol concentration. An unblinded staff will have no communication of results to any blinded study personnel during the study assessments. Blinded staff will not have access to participants' BAC results until all study assessments are complete before the checkout procedure begins.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Treatment A - 5 mg Δ9-THC + Placebo beverage (Experimental): Subjects in this arm will receive one 5 mg oral dose of THC and a placebo beverage
  Interventions: Drug: 5 mg Dronabinol (Marinol®) + Placebo Beverage
- Treatment B - 10 mg Δ9-THC + Placebo beverage (Experimental): Subjects in this arm will receive one 10 mg oral dose of THC and a placebo beverage
  Interventions: Drug: 10 mg Dronabinol (Marinol®) + Placebo Beverage
- Treatment C - 5 mg Δ9-THC + Alcohol beverage with BAC target of 0.08% (Experimental): Subjects in this arm will receive one 5 mg oral dose of THC and an alcohol beverage targeting a blood alcohol concentration (BAC) of 0.08%
  Interventions: Drug: 5 mg Dronabinol (Marinol®) + Alcohol Beverage
- Treatment D - 10 mg Δ9-THC + Alcohol beverage with BAC target of 0.08% (Experimental): Subjects in this arm will receive one 10 mg oral dose of THC and an alcohol beverage targeting a blood alcohol concentration (BAC) of 0.08%
  Interventions: Drug: 10 mg Dronabinol (Marinol®) + Alcohol Beverage
- Treatment E - Placebo capsule + Alcohol beverage with BAC target of 0.08% (Active Comparator): Subjects in this arm will receive one placebo capsule and an alcohol beverage targeting a blood alcohol concentration (BAC) of 0.08% as a positive control
  Interventions: Drug: Placebo Capsule + Alcohol Beverage
- Treatment F - Placebo capsule + Placebo beverage (Placebo Comparator): Subjects in this arm will receive one placebo capsule and a placebo beverage
  Interventions: Drug: Placebo Capsule + Placebo Beverage

INTERVENTIONS:
Drug: 5 mg Dronabinol (Marinol®) + Placebo Beverage — Subjects in this arm will receive one dose of 5 mg THC (Dronabinol) with a placebo beverage in one of the assigned treatment days.
  Arms: Treatment A - 5 mg Δ9-THC + Placebo beverage
Drug: 10 mg Dronabinol (Marinol®) + Placebo Beverage — Subjects in this arm will receive one dose of 10 mg THC (Dronabinol) with a placebo beverage in one of the assigned treatment days.
  Arms: Treatment B - 10 mg Δ9-THC + Placebo beverage
Drug: 5 mg Dronabinol (Marinol®) + Alcohol Beverage — Subjects in this arm will receive one dose of 5 mg THC (Dronabinol) with an alcoholic beverage (to achieve a target BAC of 0.08%) in one of the assigned treatment days.
  Arms: Treatment C - 5 mg Δ9-THC + Alcohol beverage with BAC target of 0.08%
Drug: 10 mg Dronabinol (Marinol®) + Alcohol Beverage — Subjects in this arm will receive one dose of 10 mg THC (Dronabinol) with an alcoholic beverage (to achieve a target BAC of 0.08%) in one of the assigned treatment days.
  Arms: Treatment D - 10 mg Δ9-THC + Alcohol beverage with BAC target of 0.08%
Drug: Placebo Capsule + Alcohol Beverage — Subjects in this arm will receive placebo capsule with an alcoholic beverage (to achieve a target BAC of 0.08%) in one of the assigned treatment days.
  Arms: Treatment E - Placebo capsule + Alcohol beverage with BAC target of 0.08%
Drug: Placebo Capsule + Placebo Beverage — Subjects in this arm will receive a placebo capsule with a placebo beverage in one of the assigned treatment days.
  Arms: Treatment F - Placebo capsule + Placebo beverage

SUMMARY:
With the increasing prevalence and use of cannabis products by the public, there exists a need to better understand the safety impact of cannabis use, particularly when it comes to subjective perceptions of drug effect and driving impairment. This study aims to evaluate the dose-dependent effects of oral Δ9-THC alone and in combination with alcohol (0.08% BAC [Blood Alcohol Concentration]) on driving performance and subjective feeling in healthy adults. The results of this study will address current knowledge gaps on the effects of oral Δ9-THC on driving impairment across a clinically relevant dose range.

DETAILED DESCRIPTION:
The cannabis plant contains bioactive compounds known as cannabinoids, with delta-9 tetrahydrocannabidiol (Δ9-THC) and cannabidiol (CBD) being the most well-known cannabinoids in varieties of cannabis. With the increasing prevalence and use of cannabis products by the public, there exists a need to better understand the safety impact of cannabis use, particularly when it comes to subjective perceptions of drug effect and driving impairment. Studies have evaluated the effects of Δ9-THC on perception and driving capacity, however they have largely focused on inhaled routes of administration in experienced users and at relatively high doses. Research on the impact of oral Δ9-THC use in occasional users at lower doses (10 mg and below) on driving capacity is limited. Furthermore, despite the increasing prevalence of concurrent cannabis and alcohol use, there also remains a significant gap in research examining the combined effects of oral THC and alcohol on driving performance. This study aims to evaluate the dose-dependent effects of oral Δ9-THC alone and in combination with alcohol (0.08% BAC [Blood Alcohol Concentration]) on driving performance and subjective feeling in healthy adults. These effects will also be compared to the established alcohol-related impairment benchmark of blood alcohol content (0.08% BAC). The inclusion of an alcohol-only arm targeting 0.08% BAC will serve as a relevant positive control, representing the legal intoxication threshold in most states in the USA and providing a well-characterized impairment baseline against which THC and THC/alcohol combination effects can be measured. The results of this study will address current knowledge gaps on the effects of oral Δ9-THC on driving impairment across a clinically relevant dose range.

In this randomized, double-blind, 6-period crossover study, 48 healthy adult volunteers with driving experience and previous cannabis exposure will receive single oral doses across six treatment conditions: 5 mg THC, 10 mg THC, 5 mg THC combined with alcohol (target BAC of 0.08%), 10 mg THC combined with alcohol (target BAC of 0.08%), alcohol alone (target BAC of 0.08%), and matched placebo, with washout periods between treatments. The study will evaluate the dose-dependent effects of Δ9-THC (with and without alcohol) on both objective driving performance and subjective participant experience. Objectives primarily include standardized driving simulator assessments measuring standard deviation of lateral position (SDLP) and standard deviation of speed (SDSP), as well as subjective effects measured through use of Visual Analogue Scales (VAS). Assessments will be conducted at baseline and predetermined intervals post-dose over 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Subject signs an IRB approved written informed consent and privacy language as per national regulations (e.g., Health Insurance Portability and Accountability Act authorization) before any study related procedures are performed.
2. Subject is a healthy, non-smoking man or woman, 21 to 55 years of age, inclusive, who weighs at least 50 kg (110 lbs) and has a body mass index of 18.5 to 33.0 kg/m2, inclusive, at Screening and check-in (Day -1).
3. Subject possesses a valid U.S. driver's license and has driven a minimum of 600 miles per year for the previous 3 years.
4. During screening subjects will be assessed using a driving simulation test. Subject must not demonstrate any motion sickness as determined by the investigator and defined in the driving simulation operations manual and subject must not have erratic driving as defined in the Screening Visit Driving Practice Assessment Operational Manual.
5. Subject has normal medical history findings, clinical laboratory results, vital sign measurements, 12-lead ECG results, and physical examination findings at screening and check-ins or, if abnormal, the abnormality is not considered clinically significant (as determined and documented by the investigator or designee). Out of range tests may be repeated once for confirmation at screening and/or check-ins at investigator's discretion.
6. Subject is an occasional user of cannabis, defined as having at least one cannabis exposure within the last 6 months, but no daily use pattern and no cannabis exposure within the past month.
7. Subject has consumed alcohol equivalent to achieving approximately 0.10% BAC (approximately 3-4 standard drinks for females and 4-5 drinks for males over 1-2 hours) within the past year without experiencing significant adverse reactions. (Note: 1 standard drink = 12 ounces of beer [5% alcohol by volume], 5 ounces of wine [12% alcohol by volume], or 1.5 ounce of distilled spirits [40% alcohol]).
8. Subject must report at least 1 instance of simultaneous alcohol and cannabis use over the past one year without experiencing significant adverse reactions based on investigator discretion.
9. Participants must agree to refrain from using any of the following for the duration of the study: alcohol, nicotine containing products, marijuana (except for provided study drug) or marijuana-derived products, hemp or hemp-derived products, including CBD, and illicit drugs of any kind. Only THC and alcohol administered at the study site will be permitted.
10. Subject must test negative for severe acute respiratory syndrome corona virus 2 (SARS-CoV-2) by a rapid antigen test at check-in. If a subject's test comes back as invalid, the test can be repeated.
11. Female subjects must be of non-childbearing potential (non-childbearing potential includes post-menopausal females defined as spontaneous amenorrhea for at least 12 months with FSH in the post-menopausal range or females who have undergone a surgical procedure that prevents pregnancy (e.g., hysterectomy, bilateral tubal ligation, occlusion, or salpingo-oophorectomy) or, if they are of childbearing potential, they must have negative serum HCG at screening and check-in and be practicing 2 effective methods of birth control (as determined by the investigator or designee; only one of the methods, but not both, may be a barrier technique) from Screening until at least 3 months after the end of the study. They must agree not to donate eggs for 30 days until after study completion.
12. Male subjects must agree to practice 2 effective methods of birth control (as determined by the investigator or designee) beginning at check-in (Day -1) until at least 3 months after the last dose of study drug. Subject must also agree to inform female partner(s) about participation in the study and ensure they are using a highly effective form of contraception (e.g., hormonal birth control or copper IUD). Male subjects may not donate sperm for 90 days after the end of the study.
13. Subject agrees to and is highly likely (as determined by the investigator) to comply with the protocol defined procedures and to complete the study.

Exclusion Criteria:

1. A history of cannabis use disorder or use of any psychoactive drug in the last month.
2. Any reported history of alcohol intolerance.
3. Alcohol intolerance as detected by ethanol patch testing.
4. Subject has a dry mouth or history of salivary gland disfunction or surgery.
5. A history of any psychiatric diagnosis, including mood, anxiety, and psychotic disorders.
6. Any family history of schizophrenia or other psychotic illness.
7. Any history of seizures, epilepsy, or traumatic brain injury.
8. History of syncope within 3 months prior to screening or any history of recurrent and/or unexplained episodes of syncope.
9. A positive test result for alcohol and drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, alcohol, opiates, phencyclidine, propoxyphene, methadone, ) at screening and check-in (Day -1).
10. Use or intend to use any medications other than birth control, including prescription, OTC, herbal or recreational products (excluding cannabis) in the 14 days prior to check-in (Day -1), unless deemed acceptable by the investigator.
11. Currently participating in another clinical study of an investigational drug or has been treated with any investigational drug within 30 days or 5 half-lives (whichever is longer) of dosing for this study.
12. Subject has used nicotine-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff, electronic cigarettes) within 6 weeks of Screening. Subjects must refrain from using these throughout the study.
13. Subject is unable to tolerate a controlled, quiet study conduct environment, including avoidance of music, television, movies, games, and activities that may cause excitement, emotional tension, or arousal during the prespecified time points.
14. Subject has known or suspected allergies or sensitivities to the study drug, delta 9-THC or sesame seeds/oil.
15. Subject has a history of consuming more than 14 units of alcoholic beverages per week within 6 months before Screening, has a history of alcohol use disorder or drug/chemical/substance abuse within 2 years before Screening (Note: 1 unit = 12 ounces of beer, 5 ounces of wine, or 1.5 ounce of spirits/hard liquor).
16. Subject tests positive for potential active alcohol use disorder (as determined by a score of 3 or greater on the Alcohol Use Disorders Identification Test-Consumption (AUDIT-C).
17. Subject has a history of suicidal ideation or previous suicide attempts.
18. Subject has a history or evidence of a clinically significant disorder, condition, or disease (e.g., cancer, human immunodeficiency virus [HIV], hepatic or renal impairment) that, in the opinion of the investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.
19. Subject has a diagnosis of COVID-19 or any signs or symptoms that are consistent with COVID-19 per CDC recommendations at screening or check-in (Day -1). These include subjects with fever or chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, diarrhea, or other symptoms indicative of likely COVID-19 in the opinion of the investigator.
20. Subject has any condition possibly affecting study drug absorption (e.g., gastrectomy, Crohn's disease, irritable bowel syndrome).
21. Subject has clinical laboratory test results (hematology, serum chemistry and urinalysis) at screening or check-ins that are outside the reference ranges provided by the clinical laboratory and considered clinically significant by the investigator. Out of range tests may be repeated once for confirmation at screening and/or check-ins at investigator's discretion.
22. Subject has a mean systolic blood pressure <90 or >140 mmHg or a mean diastolic blood pressure <50 or >90 mmHg at either screening or check-ins, unless determined not clinically significant per investigator. Blood pressure will be measured after the subject has been resting in a sitting position for approximately 5 minutes. Two blood pressure repeats will be permitted in instances where initial measures out of normal range.
23. Subject has a positive test result at screening for HIV 1 or 2 antibody, hepatitis C virus antibodies, or hepatitis B surface antigen.
24. Subject is unable or unwilling to undergo multiple venipunctures for blood sample collection because of poor tolerability or is unlikely to complete the study due to poor venous access.
25. Subject has had any significant blood loss, donated 1 unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days, or donated plasma within 7 days before check-in.
26. Subject with any visual or hearing impairment that will prevent accurate completion of study assessments (as determined by the investigator).
27. Subject has any other condition that precludes his or her participation in the study (as determined by the investigator).

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2026-04-14 (Estimated); Study Completion 2026-04-14 (Estimated)

PRIMARY OUTCOMES:
Simulated driving performance as measured by Standard Deviation of Lateral Position (SDLP) after Δ9-THC administration alone or in combination with alcohol compared to alcohol alone. | Up to 8 hours after study drug administration.
  Simulated driving performance will be measured by the endpoint standard deviation of lateral position (SDLP) using a STISIM (model M4000-R) driving simulator after Δ9-THC administration (5 mg, 10 mg, 5 mg with alcohol, 10 mg with alcohol) compared to active control (alcohol alone).

SECONDARY OUTCOMES:
Simulated driving performance as measured by Standard Deviation of Lateral Position (SDLP) after Δ9-THC administration alone or in combination with alcohol compared to placebo. | Up to 8 hours after study drug administration.
  Simulated driving performance will be measured by the endpoint standard deviation of lateral position (SDLP) using a STISIM (model M4000-R) driving simulator after Δ9-THC administration (5 mg, 10 mg, 5 mg with alcohol, 10 mg with alcohol) compared to placebo.
Simulated driving performance as measured by Standard Deviation of Speed Position (SDSP) after Δ9-THC administration alone or in combination with alcohol compared to placebo. | Up to 8 hours after study drug administration.
  Simulated driving performance will be measured by the endpoint standard deviation of speed position (SDSP) using a STISIM (model M4000-R) driving simulator after Δ9-THC administration (5 mg, 10 mg, 5 mg with alcohol, 10 mg with alcohol) compared to placebo.
Simulated driving performance as measured by Standard Deviation of Speed Position (SDSP) after Δ9-THC administration alone or in combination with alcohol compared to alcohol alone. | Up to 8 hours after study drug administration.
  Simulated driving performance will be measured by the endpoint standard deviation of speed position (SDSP) using a STISIM (model M4000-R) driving simulator after Δ9-THC administration (5 mg, 10 mg, 5 mg with alcohol, 10 mg with alcohol) compared to alcohol alone.
Maximum subjective self-rated driving impairment after Δ9-THC administration alone or in combination with alcohol compared to placebo. | Up to 24 hours after study drug administration.
  Maximum subjective self-rated driving impairment after Δ9-THC administration (5 mg, 10 mg, 5 mg with alcohol, 10 mg with alcohol) compared to placebo will be measured by the VAS question (VAS "drug driving impairment"): "How much did the study drug affect your driving?"
Maximum subjective feeling state of VAS "Drug Effect" after Δ9-THC administration alone or in combination with alcohol compared to placebo. | Up to 24 hours after study drug administration.
  Maximum subjective feeling state of VAS "Drug Effect" after Δ9-THC administration (5 mg, 10 mg, 5 mg with alcohol, 10 mg with alcohol) compared to placebo will be measured by the VAS question (VAS "Drug Effect"): "Are you feeling a drug effect right now?"
Maximum subjective feeling state of VAS "Willingness to Drive" after Δ9-THC administration alone or in combination with alcohol compared to placebo. | Up to 24 hours after study drug administration.
  Maximum subjective feeling state of VAS "Willingness to Drive" after Δ9-THC administration (5 mg, 10 mg, 5 mg with alcohol, 10 mg with alcohol) compared to placebo will be measured by the VAS question (VAS "Willingness to Drive"): "Would you drive in your current state right now?"
Maximum subjective feeling state of VAS "Confidence in Driving" after Δ9-THC administration alone or in combination with alcohol compared to placebo. | Up to 24 hours after study drug administration.
  Maximum subjective feeling state of VAS "Confidence in Driving" after Δ9-THC administration (5 mg, 10 mg, 5 mg with alcohol, 10 mg with alcohol) compared to placebo will be measured by the VAS question (VAS Confidence in Driving): "How confident are you in your driving ability?"
Maximum subjective feeling state of VAS "Liking" after Δ9-THC administration alone or in combination with alcohol compared to placebo. | Up to 24 hours after study drug administration.
  Maximum subjective feeling state of VAS "Liking" after Δ9-THC administration (5 mg, 10 mg, 5 mg with alcohol, 10 mg with alcohol) compared to placebo will be measured by the VAS question (VAS Liking): "How much do you like the drug effects right now?"
Maximum subjective feeling state of VAS "High" after Δ9-THC administration alone or in combination with alcohol compared to placebo. | Up to 24 hours after study drug administration.
  Maximum subjective feeling state of VAS "High" after Δ9-THC administration (5 mg, 10 mg, 5 mg with alcohol, 10 mg with alcohol) compared to placebo will be measured by the VAS question (VAS High): "How high do you feel right now?"
Maximum subjective feeling state of VAS "Bad Effects" after Δ9-THC administration alone or in combination with alcohol compared to placebo. | Up to 24 hours after study drug administration.
  Maximum subjective feeling state of VAS "Bad Effects" after Δ9-THC administration (5 mg, 10 mg, 5 mg with alcohol, 10 mg with alcohol) compared to placebo will be measured by the VAS question (VAS Bad Effects): "Are you feeling any bad effects right now?"
Maximum subjective feeling state of VAS "Drowsy" after Δ9-THC administration alone or in combination with alcohol compared to placebo. | Up to 24 hours after study drug administration.
  Maximum subjective feeling state of VAS "Drowsy" after Δ9-THC administration (5 mg, 10 mg, 5 mg with alcohol, 10 mg with alcohol) compared to placebo will be measured by the VAS question (VAS Drowsy): "How drowsy do you feel right now?"
Maximum subjective feeling state of VAS "Take Drug Again" after Δ9-THC administration alone or in combination with alcohol compared to placebo. | Up to 24 hours after study drug administration.
  Maximum subjective feeling state of VAS "Take Drug Again" after Δ9-THC administration (5 mg, 10 mg, 5 mg with alcohol, 10 mg with alcohol) compared to placebo will be measured by the VAS question (VAS Take Drug Again): "How likely are you to take this drug again?"

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Fein, MD, Principal Investigator — Spaulding Clinical Research LLC
Locations (2):
- United States (2):
  - Spaulding Clinical Research, West Bend, Wisconsin
  - Spaulding Clinical, West Bend, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Plan is to make data from the study publicly available as part of a manuscript publication. In addition, the protocol and statistical analysis plan will be made available online at this site as well as with any eventual publications.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available at the time of manuscript publication.
Access Criteria: No restrictions

REFERENCES:
- [Background] Cleveland Clinic. Blood Alcohol Content (BAC). https://my.clevelandclinic.org/health/diagnostics/22689-blood-alcohol-content-bac
- [Background] Dronabinol (Marinol®) capsule label obtained from https://www.accessdata.fda.gov/drugsatfda_docs/label/2023/018651s033lbl.pdf
- [Background] Zamarripa CA, Novak MD, Weerts EM, Vandrey R, Spindle TR. The effects of oral and vaporized cannabis alone, and in combination with alcohol, on driving performance using the STISIM driving simulator: A two-part, double-blind, double-dummy, placebo-controlled, randomized crossover clinical laboratory protocol. Front Pharmacol. 2022 Sep 6;13:964749. doi: 10.3389/fphar.2022.964749. eCollection 2022. PMID 36147331
- [Background] Garrisson H, Scholey A, Verster JC, Shiferaw B, Benson S. Effects of alcohol intoxication on driving performance, confidence in driving ability, and psychomotor function: a randomized, double-blind, placebo-controlled study. Psychopharmacology (Berl). 2022 Dec;239(12):3893-3902. doi: 10.1007/s00213-022-06260-z. Epub 2022 Nov 2. PMID 36322184
- [Background] Weerts EM, Wand GS, Maher B, Xu X, Stephens MA, Yang X, McCaul ME. Independent and Interactive Effects of OPRM1 and DAT1 Polymorphisms on Alcohol Consumption and Subjective Responses in Social Drinkers. Alcohol Clin Exp Res. 2017 Jun;41(6):1093-1104. doi: 10.1111/acer.13384. Epub 2017 Apr 26. PMID 28376280
- [Background] Fisher HR, Simpson RI, Kapur BM. Calculation of blood alcohol concentration (BAC) by sex, weight, number of drinks and time. Can J Public Health. 1987 Sep-Oct;78(5):300-4. No abstract available. PMID 3690446
- [Background] Veldstra JL, Bosker WM, de Waard D, Ramaekers JG, Brookhuis KA. Comparing treatment effects of oral THC on simulated and on-the-road driving performance: testing the validity of driving simulator drug research. Psychopharmacology (Berl). 2015 Aug;232(16):2911-9. doi: 10.1007/s00213-015-3927-9. Epub 2015 May 10. PMID 25957748
- [Background] Brooks-Russell A, Brown T, Friedman K, Wrobel J, Schwarz J, Dooley G, Ryall KA, Steinhart B, Amioka E, Milavetz G, Sam Wang G, Kosnett MJ. Simulated driving performance among daily and occasional cannabis users. Accid Anal Prev. 2021 Sep;160:106326. doi: 10.1016/j.aap.2021.106326. Epub 2021 Aug 14. PMID 34403895
- [Background] Hartman RL, Huestis MA. Cannabis effects on driving skills. Clin Chem. 2013 Mar;59(3):478-92. doi: 10.1373/clinchem.2012.194381. Epub 2012 Dec 7. PMID 23220273
- [Background] Bosker WM, Kuypers KP, Theunissen EL, Surinx A, Blankespoor RJ, Skopp G, Jeffery WK, Walls HC, van Leeuwen CJ, Ramaekers JG. Medicinal Delta(9) -tetrahydrocannabinol (dronabinol) impairs on-the-road driving performance of occasional and heavy cannabis users but is not detected in Standard Field Sobriety Tests. Addiction. 2012 Oct;107(10):1837-44. doi: 10.1111/j.1360-0443.2012.03928.x. Epub 2012 Jul 12. PMID 22553980
- [Background] Schnakenberg Martin AM, Flynn LT, Sefik E, Luddy C, Cortes-Briones J, Skosnik PD, Pittman B, Ranganathan M, D'Souza DC. Preliminary study of the interactive effects of THC and ethanol on self-reported ability and simulated driving, subjective effects, and cardiovascular responses. Psychopharmacology (Berl). 2023 Jun;240(6):1235-1246. doi: 10.1007/s00213-023-06356-0. Epub 2023 Apr 12. PMID 37045988
- [Background] Manning B, Hayley AC, Catchlove S, Shiferaw B, Stough C, Downey LA. Effect of CannEpil(R) on simulated driving performance and co-monitoring of ocular activity: A randomised controlled trial. J Psychopharmacol. 2023 May;37(5):472-483. doi: 10.1177/02698811231170360. Epub 2023 May 2. PMID 37129083
- [Background] Hartman RL, Brown TL, Milavetz G, Spurgin A, Pierce RS, Gorelick DA, Gaffney G, Huestis MA. Cannabis effects on driving lateral control with and without alcohol. Drug Alcohol Depend. 2015 Sep 1;154:25-37. doi: 10.1016/j.drugalcdep.2015.06.015. Epub 2015 Jun 23. PMID 26144593
- [Background] Hartley S, Simon N, Cardozo B, Larabi IA, Alvarez JC. Can inhaled cannabis users accurately evaluate impaired driving ability? A randomized controlled trial. Front Public Health. 2023 Nov 22;11:1234765. doi: 10.3389/fpubh.2023.1234765. eCollection 2023. PMID 38074719
- [Background] Arkell TR, Vinckenbosch F, Kevin RC, Theunissen EL, McGregor IS, Ramaekers JG. Effect of Cannabidiol and Delta9-Tetrahydrocannabinol on Driving Performance: A Randomized Clinical Trial. JAMA. 2020 Dec 1;324(21):2177-2186. doi: 10.1001/jama.2020.21218. PMID 33258890